CLINICAL TRIAL: NCT01002287
Title: An Evaluation of the SprayShield Adhesion Barrier System in Reducing Post-Operative Adhesion in Abdominal Surgery
Brief Title: An Evaluation of SprayShield in Reducing Post-Operative Adhesion Formation Following Major Open Abdominal Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated for business purposes, not for safety or efficacy reasons.
Sponsor: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ABD-08-001
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Results first posted 2014-01-29 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Ulcerative Colitis; Familial Polyposis
MeSH Terms: conditions — Colitis, Ulcerative; Adenomatous Polyposis Coli

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- SprayShield Adhesion Barrier (Experimental): SprayShield Adhesion Barrier
  Interventions: Device: SprayShield Adhesion Barrier System
- Control (Sham Comparator): Good Surgical Technique Alone
  Interventions: Procedure: Good Surgical Technique Alone

INTERVENTIONS:
Device: SprayShield Adhesion Barrier System — Adhesion Barrier Device
  Arms: SprayShield Adhesion Barrier
Procedure: Good Surgical Technique Alone — Good Surgical Technique Alone
  Arms: Control

SUMMARY:
This will be a prospective, multi-center, randomized, single blind study to collect and evaluate post-market clinical data on the SprayShield Adhesion Barrier System as an adjuvant to good surgical technique for the reduction of postoperative adhesion formation following major open abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ulcerative colitis or familial polyposis and require two-stage surgery for treatment of either of these disorders will be eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-10; Primary Completion 2010-10 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Covidien, Bedford, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Initiation: 31October2009 Study Termination: 24March2010
  Study was conducted in hospitals.
Groups:
- SprayShield Adhesion Barrier: SprayShield Adhesion Barrier + Good Surgical Technique
Period: Overall Study
Arm/Group | SprayShield Adhesion Barrier | Control
Started | 8 | 3
Completed | 8 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SprayShield Adhesion Barrier | Control | Total
Number analyzed (Participants) | 8 | 3 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 3 | 10
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.5 (12.6) | 37.7 (19.8) | 45.5 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 5 | 3 | 8
Region of Enrollment [Number; unit: participants]
  Czech Republic | 3 | 2 | 5
  Poland | 5 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of Adhesions, Defined as the Proportion of Subjects Presenting at the Follow-up Surgery (10-12 Weeks) With One or More Adhesions to the Midline Incision, Regardless of Extent and/or Severity.
Time Frame: 10-12 Weeks post Initial Surgery for J-Pouch
Population: All 11 patients met the per protocol population requirements specified in the protocol and statistical analysis plan.
Measure: Number; unit: percentage of subjects with adhesions
Arm/Group | SprayShield Adhesion Barrier | Control
Number analyzed (Participants) | 8 | 3
percentage of subjects with adhesions | 37.5 | 66.7

2. Secondary Outcome: Severity of Adhesions
Description: Worst midline adhesion severity score. The severity of adhesions was categorized as filmy thickness, avascular; moderate thickness, limited vascularity; and dense thickness, vascularised. The corresponding numeric severity ratings are "1", "2", and "3". Subjects without adhesions were assigned a severity rating of "0".
Time Frame: Average 10-12 weeks post surgery
Population: All 11 subjects met the definition of per protocol population in the protocol and statistical analysis plan.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SprayShield Adhesion Barrier | Control
Number analyzed (Participants) | 8 | 3
units on a scale | 0.9 (1.2) | 1.3 (1.2)

3. Secondary Outcome: Adhesion Involvement Along the Midline Incision (Percentage)
Description: The proportion of the total length of the initial midline incision associated with any adhesion at the time of the follow-up surgery, as determined by dividing the length of the incision associated with adhesions (cm) by the overall initial midline incision length (cm). This calculates the extent of adhesion involvement as a percentage.
Time Frame: average 10-12 weeks post surgery
Population: These patients must have values for length of the incision associated with adhesions (cm) and for length of initial midline incision (cm) in order to calculate Extent of Adhesion Involvement (%). NOTE: Extent of Adhesion Involvement (%) = length of the incision associated with adhesions (cm) / length of initial midline incision (cm) * 100.
Measure: Mean (Standard Deviation); unit: percentage of midline incision
Arm/Group | SprayShield Adhesion Barrier | Control
Number analyzed (Participants) | 1 | 2
percentage of midline incision | 66.7 (0) | 76.3 (33.5)

4. Secondary Outcome: Mobilization Time
Description: The time (minute) required to incise and mobilize the ileal loop in preparation for reanastomosis for ileostomy closure.
Time Frame: average 10-12 weeks post surgery
Population: All 11 patients meet the per protocol population defined in the protocol and the statistical analysis plan.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | SprayShield Adhesion Barrier | Control
Number analyzed (Participants) | 8 | 3
minutes | 41.0 (13.7) | 43.3 (2.9)

ADVERSE EVENTS:
Arm/Group | SprayShield Adhesion Barrier | Control
Serious Adverse Events (participants affected / at risk) | 2/8 | 1/3
Other Adverse Events (participants affected / at risk) | 4/8 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SprayShield Adhesion Barrier (N=8) | Control (N=3)
Fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Surgical Skin Tear (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SprayShield Adhesion Barrier (N=8) | Control (N=3)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Impaired Healing (General disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No